CLINICAL TRIAL: NCT04787042
Title: A First-In-Human Phase 1/2 Open-Label Study of Intravenous ST-067, Subcutaneous ST-067 with or Without Obinutuzumab Pre-Treatment, and ST-067 in Combination with Pembrolizumab in Subjects with Advanced Solid Malignancies
Brief Title: Phase 1a and Phase 2 Study for Safety, Preliminary Efficacy, PK and PD of ST-067
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Simcha IL-18, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ST-067-001; KEYNOTE-E64 (Other: Merck); MK-3475-E64 (Other: Merck)
Record Dates: First submitted 2021-02-16; First posted 2021-03-08 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Solid Tumor; Melanoma; Renal Cell Carcinoma; Triple-negative Breast Cancer; Non Small Cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck; Carcinoma; MSI-High
MeSH Terms: conditions — Neoplasms; Melanoma; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Carcinoma | interventions — obinutuzumab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Dose escalation and expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase 1a, Dose Escalation (Experimental): In the Phase 1a monotherapy study, the starting dose of ST-067 will be 30 μg/kg, with a total of 7 dose level cohorts planned.
  The starting dose for the IV infusion monotherapy dosing will be 60 µg/kg.
  Patients will be treated every week with ST-067 in all cohorts. The DLT period is 28 days after the initial dose of ST-067. According to the mTPI schema initially there will be 3 patients per cohort until the first DLT is observed at which point cohorts will be expanded according to the predetermined mTPI design. Up to 12 patients will be treated at the RP2D.
  Interventions: Biological: ST-067
- Phase 2, Expansion (Experimental): Phase 2 will enroll patients aged 18 years or older diagnosed with the following solid tumors: melanoma, renal cell carcinoma (RCC), triple negative breast cancer (TNBC), non-small cell lung cancer (NSCLC), squamous cell carcinoma of the head and neck (SCCHN), and microsatellite instability-high (MSI-Hi) tumors at the RP2D.
  Interventions: Biological: ST-067
- Phase 1a, Dose Escalation, ST-067 SC + Obinutuzumab Pre-treatment (Experimental): Patients will be treated every week with ST-067 in all cohorts. The DLT period is 28 days after the initial dose of ST-067. According to the mTPI schema initially there will be 3 patients per cohort until the first DLT is observed at which point cohorts will be expanded according to the predetermined mTPI design.
  The starting dose for ST-067 with obinutuzumab pre-treatment will be 120µg/kg. Obinutuzumab will be administered at 1000 mg daily via IV infusion on 2 consecutive days, with the first dose given at least 7 days prior to first dose of SC ST-067.
  Interventions: Biological: ST-067; Biological: Obinutuzumab 25 MG/1 ML Intravenous Solution [GAZYVA]
- Phase 1 combination therapy (Experimental): Phase 1 dose escalation in combination with pembrolizumab will start at a dose of 30 µg/kg of ST-067 and 200 mg every 3 weeks of pembrolizumab. Patients will be treated every week with ST-067 and every three weeks with pembrolizumab. The MTD will be determined based on the mTPI design.
  Interventions: Biological: ST-067; Biological: pembrolizumab

INTERVENTIONS:
Biological: ST-067 — ST-067 is an engineered variant of human interleukin-18.
Biological: Obinutuzumab 25 MG/1 ML Intravenous Solution [GAZYVA] — Obinutuzumab is a humanized anti-CD20 monoclonal antibody of the IgG1 subclass. It recognizes a specific epitope of the CD20 molecule found on B-cells.
  Other Names: GAZYVA
  Arms: Phase 1a, Dose Escalation, ST-067 SC + Obinutuzumab Pre-treatment
Biological: pembrolizumab — Pembrolizumab is a potent humanized immunoglobulin G4 monoclonal antibody.
  Other Names: KEYTRUDA®
  Arms: Phase 1 combination therapy

SUMMARY:
This is a multiphase, multicenter study, which includes a Phase 1a open-label, dose escalation monotherapy study of ST-067 given as an SC injection with or without obinutuzumab [Gazyva®] pre-treatment, by IV infusion, and in combination with pembrolizumab. A Phase 2 monotherapy arm is also planned; the exact design of the Phase 2 study elements with respect to formulation and pre-treatment will be determined after completion of the Phase 1 study portion of the trial.

DETAILED DESCRIPTION:
Phase 1a is designed to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of ST067, administered by subcutaneous (SC) or intravenous (IV) dosing, in subjects with relapsed or refractory solid tumors, as well as to determine the MTD and recommended Phase 2 dose of ST067, administered SC with obinutuzumab (Gazyva®) as pretreatment in subjects with relapsed or refractory solid tumors using a modified toxicity probability interval (mTPI) design. There will be evaluations of ST-067 PK and PD effects.

Phase 2 will evaluate the preliminary efficacy of ST-067 administered at the RP2D to patients with the following tumor types. A Simon 2 stage design is used to calculate the sample size and early stopping rules will be employed in the event of lack of efficacy in any of the cohorts. RECIST 1.1 will be used to assess tumor response every 8-12 weeks.

* Melanoma (n=28)
* Renal cell carcinoma (n=25)
* Triple-negative best cancer (n=25)
* Non-small cell lung cancer (n=25)
* squamous cell carcinoma of the head and neck (n=28)
* MSI-Hi tumors (n=25)

A Simon 2 stage design is used to calculate the sample size and early stopping rules will be employed in the event of lack of efficacy in any of the cohorts. RECIST 1.1 will be used to assess tumor response every 8-12 weeks.

Safety will be assessed for each patient throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥18 years
2. Must provide written informed consent and any authorizations required by local law
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Have histologically or cytologically confirmed diagnosis of advanced/metastatic solid tumor

   For Phase 1a, the following solid tumors are allowed: Melanoma, Merkel cell, RCC, urothelial, NSCLC,TNBC, SCCHN, microsatellite instability high, high tumor mutation burden (Hi TMB) or mismatch repair deficient, gastric, cervical, endometrial, cutaneous squamous, small cell lung, esophageal, hepatocellular carcinoma and platinum resistant ovarian cancer.
   1. For patients who have developed disease progression through standard therapy, or
   2. For patients whom standard of care therapy that prolongs survival is unavailable or unsuitable (according to the investigator and after consultation with the Medical Monitor) For Phase 1 combination therapy dose escalation, the following solid tumors are allowed: Melanoma, Merkel cell, RCC, urothelial, NSCLC (with no EGFR, TRK receptor, or ALK positive mutations/fusions), TNBC, SCCHN, MSI-Hi tumors, Hi TMB or mismatch repair deficient, gastric, cervical, endometrial, cutaneous squamous, small cell lung, esophageal, and HCC

      * TNBC is diagnosed in a tumor which does not express estrogen receptor or progesterone receptor, is not human epidermal growth factor receptor 2 (HER2) 3+ on IHC or is negative by fluorescence in situ hybridization (FISH).
      * MSI high tumor should have mutations in 30% or more microsatellites by PCR or be negative for MSH1/2/6 or PMS-2 by IHC.
      * Hi-TMB high tumor has 10 mut/Mb or greater calculated from whole genome sequencing or whole exome sequencing

   For Phase 2, the following solid tumors are allowed:

   Melanoma, RCC, TNBC, NSCLC, SCCHN, and MSI-Hi tumors
5. Has at least 1 measurable lesion per RECIST 1.1 criteria which has not been biopsied or received prior irradiation
6. Has an accessible tumor for biopsy pre- and on-treatment (mandatory).

Exclusion Criteria:

1. History of another malignancy
2. Known symptomatic brain metastases requiring >10 mg/day of prednisolone or equivalent
3. Significant cardiovascular disease (MI, thrombotic events,) within 6 months prior to study treatmentSignificant ECG abnormalities (Phase 1a and 2 monotherapy only) including unstable cardiac arrhythmia requiring medication, second-degree atrioventricular block type II, third degree AV
4. Any degree of respiratory compromise (from either malignant or non-malignant disease)
5. Evidence of an ongoing systemic bacterial, fungal, or viral infection
6. Has received a live vaccine within 30 days
7. Major surgery within 4 weeks
8. Prior solid organ or bone marrow progenitor cell transplantation
9. Prior high dose chemotherapy requiring stem cell rescue
10. History of active autoimmune disorders
11. Ongoing immunosuppressive therapy, including systemic or enteric corticosteroids.
12. Treatment with an approved, systemic anticancer therapy or an investigational agent within 4 weeks of Day 1
13. A positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) viral test within 28 days prior to dosing, unless there is Investigator-confirmed clinical recovery on or before C1D1
14. Subjects with adrenal insufficiency
15. Subjects with any chemistry or hematology laboratory values that are ≥Grade 2

    Additional exclusion criteria for Phase 1 combination therapy only:
16. Presence of known active CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging, clinically stable, and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
17. Prior radiotherapy within 2 weeks of start of study treatment or history of radiation pneumonitis.
18. Presence of an active documented autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine or insulin) is not considered a form of systemic treatment and is allowed. Subjects may use topical and/or inhaled corticosteroids. However, subjects with adrenal insufficiency on replacement doses of steroids are not allowed.
19. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX40, CD137), and was discontinued from that treatment due to a Grade 3 or higher irAE
20. Severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients. Subjects who have been retreated after such a reaction may be allowed after discussion with the Simcha Medical Monitor
21. History of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
22. Subjects that have received radiation therapy to the lung that is >30Gy within 6 months of the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of ST-067 in phase 1a monotherapy | Day 29
  Patients will be enrolled at a dose level that is predicted to be the MTD
Evaluate the overall safety and tolerability of ST-067 in combination with pembrolizumab | Day 29
  In patients experiencing insufficient response to a checkpoint inhibitor (PD-1) therapy administered alone or in combination.
Number of Participants With Treatment-Related Adverse Events | Day 29
  AE assessed by CTCAE 5.0
Initial assessment of efficacy in phase 2 | At 8 weeks
  Investigator-assessed ORR, defined as either a complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 based on computed tomography (CT) or magnetic resonance imaging (MRI) scans

SECONDARY OUTCOMES:
PK | Day 29
  Peak Plasma Concentration (Cmax)
ADA | Day 29
  Incidence of ADA to ST-067

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Barton, MD, Study Director — Simcha IL-18, Inc.
Locations (6):
- United States (6):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No